CLINICAL TRIAL: NCT07182617
Title: Assessing the Utility of a Remote Patient Monitoring Platform for Improving CPAP Adherence for Obstructive Sleep Apnea
Brief Title: MonitAir Remote Patient Monitoring Versus Standard of Care for CPAP Adherence in Obstructive Sleep Apnea
Acronym: MONITAIR-OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MonitAir (Industry)
Collaborators: BetterNight (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MONITAIR-CPAP-001
Record Dates: First submitted 2025-08-26; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: Sleep Apnea; Obstructive Sleep Apnea; OSA; CPAP; CPAP Adherence; Remote Patient Monitoring; Telehealth; Digital Health; Patient Engagement
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Patient Participation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two parallel arms: standard coaching program (SOC) versus MonitAir remote patient monitoring (RPM) platform.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of Care (SOC) Coaching (Active Comparator): Participants received the standard BetterNight coaching program for CPAP initiation and adherence. Monitoring was performed using existing systems (ResMed AirView, Philips Care Orchestrator, and the internal Clarity dashboard). Coaches contacted patients at scheduled checkpoints (10, 20, 45, 60, and 80 days) and provided support as needed to help patients meet Medicare adherence criteria.
  Interventions: Behavioral: Standard Coaching (SOC)
- MonitAir Remote Patient Monitoring (RPM) (Experimental): Participants received the standard BetterNight coaching program enhanced with the MonitAir RPM platform. MonitAir enabled weekly data reviews, automated text reminders, and at least one interactive telehealth session per month. Alerts for poor adherence, high residual AHI, or mask issues triggered outreach by coaches and escalation to physicians when needed. The goal was to improve CPAP adherence and patient satisfaction through continuous digital monitoring and engagement.
  Interventions: Behavioral: MonitAir RPM

INTERVENTIONS:
Behavioral: Standard Coaching (SOC) — Participants received BetterNight's standard CPAP coaching program. Monitoring was conducted through manufacturer platforms (ResMed AirView, Philips Care Orchestrator) and BetterNight's internal Clarity dashboard. Coaches contacted patients at scheduled checkpoints (10, 20, 45, 60, and 80 days) to provide education, support, and troubleshooting to help patients achieve Medicare adherence.
  Other Names: BetterNight Standard of Care
  Arms: Standard of Care (SOC) Coaching
Behavioral: MonitAir RPM — Participants received the standard BetterNight coaching program enhanced with the MonitAir remote patient monitoring platform. MonitAir enabled weekly reviews of CPAP usage data, automated text follow-ups, and at least one interactive telehealth visit per month. Coaches escalated issues such as poor adherence, high residual AHI, or mask leak to physicians as needed. The intervention aimed to improve CPAP adherence and patient satisfaction compared with standard care.
  Other Names: MonitAir Remote Patient Monitoring
  Arms: MonitAir Remote Patient Monitoring (RPM)

SUMMARY:
This study tested whether using the MonitAir remote patient monitoring (RPM) platform could improve adherence to continuous positive airway pressure (CPAP) therapy for patients with obstructive sleep apnea. Patients starting CPAP treatment with BetterNight were randomized to receive either standard coaching (control group) or enhanced monitoring with the MonitAir platform (intervention group). The study measured CPAP adherence at 30, 60, and 90 days, as well as patient satisfaction and other clinical outcomes.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a highly prevalent sleep disorder that is associated with hypertension, cardiovascular disease, diabetes, and impaired quality of life. Continuous positive airway pressure (CPAP) therapy is the gold standard treatment for OSA, but long-term adherence remains a significant challenge. Many patients discontinue therapy early, and overall adherence rates often fall below the thresholds required for symptom relief and insurance coverage.

Remote patient monitoring (RPM) has been successfully applied to other chronic diseases such as heart failure, diabetes, and asthma, improving both patient engagement and clinical outcomes. MonitAir is a HIPAA-compliant, FDA-registered Medical Device Data System (MDDS) designed to integrate CPAP device data with telehealth features, enabling clinicians to remotely track nightly usage, apnea-hypopnea index (AHI), and mask leak, while providing timely feedback and support to patients.

This randomized controlled trial was conducted in partnership with BetterNight, a nationwide provider of sleep services. A total of 200 patients with newly diagnosed OSA who were initiating CPAP therapy were randomized in a 1:1 ratio to receive either the standard BetterNight coaching program (standard of care arm) or the same program enhanced with the MonitAir RPM platform (intervention arm). The MonitAir arm included structured weekly data reviews, automated text messaging, monthly telehealth check-ins, and physician escalation when clinically indicated.

The primary outcome was CPAP adherence at 30, 60, and 90 days, defined according to Medicare criteria (≥4 hours of CPAP use per night for at least 70 percent of nights in a consecutive 30-day period). Secondary outcomes included patient satisfaction, time to reach CMS adherence, average nightly CPAP use, validated sleep quality questionnaires (FOSQ, PSQI, ESS), residual AHI, mask leak, mask on/off events, the number of mask refits, and study dropout rates with reasons.

Each patient participated for 90 days, and interim analysis was planned once 150 patients had been enrolled. Safety monitoring included routine tracking of typical CPAP side effects such as nasal dryness, rhinorrhea, facial irritation, or infection. Because all patients received CPAP therapy, no excess risks were anticipated between study arms; the only difference was the method of monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old
* Access to a smartphone (iOS or Android)
* Ability to engage in two-way text communication and audiovisual conferencing
* Home sleep test (HST) or polysomnogram (PSG) performed ≤90 days before randomization
* Apnea-Hypopnea Index (AHI) ≥5 (using 3% desaturation criteria)
* Prescribed and willing to initiate CPAP or APAP therapy
* Receiving a ResMed, Philips, or React CPAP device with a cellular modem
* CPAP data available to MonitAir and BetterNight

Exclusion Criteria:

* Department of Transportation (DOT) drivers
* Central sleep apnea or Cheyne-Stokes respirations (CSA/CSR) ≥10% of diagnostic study
* Central or mixed apneas ≥25% of AHI
* Use of BiPAP, BiPAP ST, ASV, AVAPS, or any other non-invasive ventilation modality
* Inability or unwillingness to participate in study activities or meet requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
CPAP adherence according to Medicare criteria | Days 30, 60, and 90 after CPAP initiation
  Percentage of patients meeting Medicare adherence criteria, defined as ≥4 hours of CPAP use per night for ≥70% of nights in a consecutive 30-day period, measured at 30, 60, and 90 days.

SECONDARY OUTCOMES:
Patient Satisfaction | Baseline, Day 30, Day 60, and Day 90 after starting CPAP
  Patient satisfaction with therapy measured using a 5-point Likert scale (1 = very dissatisfied; 5 = very satisfied). Higher scores reflect greater satisfaction. Administered via electronic survey.
Time to CMS-defined adherence | Baseline to Day 90 after starting CPAP
  Number of days required for each participant to meet CMS adherence criteria: ≥4 hours/night on ≥70% of nights in a consecutive 30-day period within the first 90 days. Lower values indicate faster adherence achievement.
Average nightly CPAP use | Day 30, Day 60, and Day 90 after starting CPAP
  Mean CPAP use in hours per night, calculated separately for all days and for days with usage, based on device-recorded data. Higher values indicate greater adherence to therapy.
Functional Outcomes of Sleep Questionnaire (FOSQ) | Baseline, Day 30, Day 60, and Day 90 after starting CPAP
  Sleep-related quality of life measured by the FOSQ-10. Total score range: 5 (worst) to 20 (best). Higher scores indicate better functional outcomes related to sleep.
Pittsburgh Sleep Quality Index (PSQI) | Baseline, Day 30, Day 60, and Day 90 after starting CPAP
  Patient-reported global sleep quality using PSQI. Total score range: 0 to 21. Higher scores indicate worse sleep quality. Administered via electronic survey.
Epworth Sleepiness Scale (ESS) | Baseline, Day 30, Day 60, and Day 90 after starting CPAP
  Daytime sleepiness measured by the ESS. Total score ranges from 0 to 24, with higher scores indicating greater daytime sleepiness.
Residual Apnea-Hypopnea Index (AHI) | Baseline and Day 90 or at Medicare adherence assessment
  Mean residual AHI (events/hour) captured from CPAP device while on therapy. AHI reflects apneas and hypopneas per hour of use. Lower values indicate better treatment effectiveness.
Mask leak | Day 30, Day 60, and Day 90 after starting CPAP
  Median mask leak (liters per minute) per participant as recorded by CPAP device. Lower values reflect better mask seal and improved therapy delivery.
Mask on/off events | Day 30, Day 60, and Day 90 after starting CPAP
  Mean number of times per night the CPAP mask is removed and reapplied, as recorded by the device. Lower values reflect better comfort and sleep continuity.
Mask refits | Up through Day 90 after starting CPAP
  Number of mask refitting events performed per participant during the study, as recorded by clinical staff. Fewer refits may reflect better initial fit and mask comfort.
Study dropout rate | Up through Day 90 after starting CPAP
  Proportion of participants who withdrew from the study. Reasons for dropout (e.g., discomfort, non-adherence, lost to follow-up) will be recorded and categorized.

CONTACTS AND LOCATIONS:
Locations (1):
- Remote, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data (IPD). Aggregate study results will be published in peer-reviewed journals and may be presented at conferences.

REFERENCES:
- Available data/document: Study Protocol: Research Protocol — https://drive.google.com/file/d/1Y8Ubu5Ie_BSDOER7_672YlAa5KttK5Wn/view?usp=sharing — https://drive.google.com/file/d/1Y8Ubu5Ie_BSDOER7_672YlAa5KttK5Wn/view?usp=sharing

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/17/NCT07182617/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/17/NCT07182617/ICF_001.pdf